CLINICAL TRIAL: NCT02665052
Title: Translating Intensive Arm Rehabilitation in Stroke to a Telerehabilitation Format
Acronym: TeleBATRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B1828-R
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Hemiparesis
Keywords: Rehabilitation; Motor Recovery; upper extremity
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Parallel: participants are randomized to one of 3 groups: delayed control, active clinic-based training or active home-based training for the initial phase of the study. The delay group is randomly assigned to receive either clinic-based or home-based training for the second phase of the study.
Who Masked: Outcomes Assessor
Masking Description: Blinded evaluator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Home-Based BATRAC (Experimental): Home-based BATRAC training will consist of 45 minutes of high intensity bilateral reaching and rest periods using the BATRAC followed by 15 minutes of video guided transition to task training (TTT). These videos will be linked from the VA MyHealtheVet site to study specific Youtube videos of the study therapist demonstrating the exercise. Asynchronous communication between the therapist and participant will be completed using the MyHealtheVet secure messaging system.
  Interventions: Device: Home-Based BATRAC plus TTT
- Lab-based BATRAC plus TTT (Experimental): Lab-based BATRAC will consist of 60 minutes of training in the lab (45 minutes using BATRAC and 15 minutes of TTT). BATRAC training will include high intensity bilateral reaching and rest periods followed by 15 minutes of therapist guided transition to task training (TTT).
  Interventions: Device: Lab-based BATRAC plus TTT
- Delayed Entry Usual Care (Placebo Comparator): Participants randomized to this group will initially serve as a control for the first 6 weeks of the study and not receive any study interventions except the protocol study evaluations in the same time intervals as those receiving active interventions. They will also receive weekly phone calls to record general activity level. After serving as a control, this group will be entered into their randomized active intervention group of either lab-based BATRAC + TTT training, or Lab-based Robot+ TTT.
  Interventions: Behavioral: Delayed Entry Usual Care

INTERVENTIONS:
Device: Home-Based BATRAC plus TTT — Home-based BATRAC training will consist of 60 minutes of training at home (45 minutes using the BATRAC and 15 minutes of TTT) using the BATRAC training will include high intensity bilateral reaching and rest periods using the BATRAC followed by 15 minutes of video guided transition to task training (TTT). These videos will be linked from the VA MyHealtheVet site to study specific Youtube videos of the study therapist demonstrating the exercise. Asynchronous communication between the therapist and participant will be completed using the MyHealtheVet secure messaging system.
  Arms: Home-Based BATRAC
Device: Lab-based BATRAC plus TTT — Lab-based BATRAC will consist of 60 minutes of training in the lab (45 minutes using BATRAC and 15 minutes of TTT). BATRAC training will include high intensity bilateral reaching and retrieving actions (pushing handles away and pulling them back) on a constrained linear track to promote maximum arm extension. This training will be followed by 15 minutes of transition to task training (TTT) with supervision and support as needed by the therapist.
  Arms: Lab-based BATRAC plus TTT
Behavioral: Delayed Entry Usual Care — Participants randomized to this group will initially serve as a control for the first 6 weeks of the study and not receive any study interventions except the protocol study evaluations in the same time intervals as those receiving active interventions and weekly phone calls to record general activity level.
  Arms: Delayed Entry Usual Care

SUMMARY:
Loss of arm use and strength are common problems after stroke that greatly affects independence in activities of daily living. Arm rehabilitation using robot-assisted repetitive task training has shown to improve motor recovery. However, this type of exercise cannot be done at home as these devices are large and expensive. This study will test whether a more portable, less costly, non-robotic repetitive training device called Bilateral Arm Training with Rhythmic Auditory Cuing (BATRAC) performed at home with a tele-rehabilitation format will lead to improvement in arm and hand use in patients with chronic stroke. The investigators plan to test the effectiveness of home based tele-rehabilitation with the BATRAC compared to a home and a clinic based approach.

DETAILED DESCRIPTION:
This is a longitudinal, single blind, randomized controlled trial with three parallel 6 week intervention arms that will be conducted over a three-year time period. After obtaining informed consent, and completing baseline testing, participants will be randomized to one of three study arms: 1) Home-based BATRAC Telerehab (HBT) + TTT, 2) Lab-based BATRAC (LBB) + TTT, and 3) Delayed Entry Usual Care. This delayed entry group will serve as a control for the initial six weeks of enrollment and NOT receive an active study intervention before randomizing to one of the two active interventions. Weekly phone calls will be conducted during this control period to record general activity (household or community) and monitor amount and intensity of arm use.

Participants will complete Home-based BATRAC training or Lab-based BATRAC training three times a week for 6-9 weeks for a total of 18 training sessions. Participants will then be asked to return for a follow-up after 8 weeks of no training. A study evaluator blinded to the intervention assignment will complete all outcome measures at baseline, training completion, and at the 8 week retention follow-up. The participants in the Home-based BATRAC telerehabilitation group will be given a VA's MyHealtheVet (www.myhealth.va.gov) website account for asynchronous communication with the therapist and to access the educational features and resources about stroke, exercise and caregiver support. The interventions are as described below.

1. Home-based BATRAC telerehabilitation: The BATRAC training platform will be used in conjunction with the VA MyHealtheVet website. This group will have a MyHealtheVet account to access the Secure Messaging Option for VA approved electronic messaging to the study therapist. The MyHealtheVet will provide asynchronous communication with the study therapist, and will store performance information entered by the participant and caregiver related to arm exercise duration, repetitions completed and distances reached. This account can be securely linked and is VA approved for use on any home device (computer, cell phone or tablet) with internet. MyHealtheVet training will be completed at the VA and at a one-time home visit with the participant and their identified caregiver to verify access, and use.

   BATRAC training will consist of 45 minutes of high intensity bilateral reaching and rest periods (see Lab-based BATRAC training details below) followed by 15 minutes of video guided Transition to Task Training (TTT). These videos will be linked from the VA MyHealtheVet site to study specific Youtube videos demonstrating the exercise. The initial training will occur in the lab setting with the therapist for BATRAC instruction and TTT exercise training. The participant and caregiver will have the opportunity ask questions and develop proficiency during this training session. For the TTT, each functional task will be presented via the MyHealtheVet Secure Messaging (SM) and linked by a URL to an instructive Youtube video clip of exercise sequencing, and level of difficulty. After completion of each exercise session the participant will complete a study report form attached to the SM. This information will be available for off-line assessment of performance by the research therapist. In cases of participant non-adherence, the therapist can contact the participant via phone to review exercise barriers and motivate the individual to participate. If necessary, the therapist could change the exercise parameters and send changes within the My HealtheVet SM.
2. Lab-based BATRAC + TTT training: Participants randomized to this group will receive 60 minutes of training in the lab (45 minutes using BATRAC and 15 minutes of TTT). The BATRAC training consists of high intensity bilateral reaching and retrieving (pushing handles away and pulling them back) on a constrained linear track to promote maximum arm extension. The track can be set at different angles in the work space. The training protocol is the same for both groups and will consist of four, 5-minute periods interspersed with 5-minute rest periods to avoid fatigue. An auditory metronome is set initially at the participant's preferred speed and for periods 1 and 3 participants move both arms simultaneously (in-phase). In periods 2 and 4 participants move both arms in alternating (antiphase) movements. A fifth bout of simultaneous arm movements will be included to reach the 45 minute training goal. Progression of the auditory cue frequency, direction of travel (pushing/pulling or in a diagonal) and distance of reach will be progressed every 2 weeks based on performance. If a progression cannot be sustained for the five-minute bouts by the end of the session, adjustments towards the previous level are made. This training will be followed by 15 minutes of transition to task training (TTT) as described below with supervision and support as needed by the therapist.

   Transition to Task Training (TTT): Each participant will receive 45 minutes of their randomized BATRAC intervention followed by 15 minutes of TTT. This training is functionally based in four domains of real-world tasks: homemaking, hygiene, feeding, and dressing. Two goal directed functional tasks are selected from the four domains every two weeks and prescribed to the individual based on severity level, general interests and goal. The task design is progressive in nature and difficulty is added by changing the parameters (movement amplitude) and demand (resistance) for increased generalization to real life challenges. Assist by the therapist or caregiver is provided to prevent compensatory movements from being re-enforced. For the home-based training, the caregiver will be instructed to provide this assistance through the initial personal training as well as have access to a set of videos for each of the tasks.
3. Delayed Entry Usual Care: Participants randomized to this group will initially serve as a control and not receive any study interventions except for the protocol study evaluations in the same time intervals as those receiving active interventions and weekly phone calls to record general activity level. After serving as a control, this group will be entered into their delayed active intervention group of either lab-based BATRAC + TTT training, or Lab-based Robot+ TTT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have a clinically defined unilateral hemiparetic stroke with radiologic exclusion of other diagnosis
* Stroke onset of at least 6 months prior to enrollment
* Present with moderate to severe arm impairment based on a Fugl-Meyer score ranging from 19-50 out of 66
* No previous experience using the BATRAC
* Ability to use and interact with the tele-rehabilitation platform according to study protocol
* Have an identified individual/caregiver to perform the TTT exercises if randomized to the Home Telerehabilitation group

Exclusion Criteria:

* Musculoskeletal diagnosis or significant arm pain that would interfere with positioning and use of the intervention (BATRAC) devices
* Cognitive impairment such that the participant is unable to understand the study requirements to answer the Evaluation to Sign Consent Form tool accurately
* Absence of a working telephone line or cell phone for telerehabilitation set-up if randomized to this group
* Enrollment in a concurrent rehabilitation study or actively receiving therapy for their stroke affected (study) arm
* Having received a botulinum toxin injection to the stroke affected (study) arm within 3 months of enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Conroy, DSc PT, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatnagar K, Bever CT, Tian J, Zhan M, Conroy SS. Comparing Home Upper Extremity Activity with Clinical Evaluations of Arm Function in Chronic Stroke. Arch Rehabil Res Clin Transl. 2020 Jun 18;2(2):100048. doi: 10.1016/j.arrct.2020.100048. PMID 33336184
- [Derived] Conroy SS, Harcum S, Keldsen L, Bever CT Jr. Novel use of existing technology: A preliminary study of patient portal use for telerehabilitation. J Telemed Telecare. 2022 Jun;28(5):380-388. doi: 10.1177/1357633X20950172. Epub 2020 Sep 1. PMID 32869689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-dwelling adults with chronic hemiparetic arm disability were recruited from the VA Maryland Health Care System, University of Maryland Medical System, and community between May 2017 and July 2019.
Pre-assignment Details: Of 63 enrolled participants, 44 were study trial participants and 19 were participant caregivers for the home-based group. Of the 44 study trial participants, 15 did not meet inclusion criteria resulting in 29 individuals randomized into the study.
Groups:
- Home-based BATRAC: Home-based BATRAC training consisted of 60 minutes of training at home (45 minutes of high intensity bilateral reaching and rest periods using the BATRAC followed by 15 minutes of video guided transition to task training (TTT)). The TTT videos were linked from the VA MyHealtheVet site to study specific Youtube videos of the study therapist demonstrating the exercise. Asynchronous communication between the therapist and participant was completed using the MyHealtheVet secure messaging system.
- Lab-based BATRAC Plus TTT: Lab-based BATRAC + TTT consisted of 60 minutes of training in the lab (45 minutes using BATRAC and 15 minutes of TTT). BATRAC training included high intensity bilateral reaching and rest periods followed by 15 minutes of therapist supervised and guided transition to task training (TTT).
- Delayed Entry Usual Care: Participants randomized to this group initially served as a control for the first 6 weeks of the study and did not receive any study interventions except the protocol study evaluations in the same time intervals as those receiving active interventions. They did receive weekly phone calls to record general activity level. After serving as a control, this group was entered into their randomized active intervention group of either lab-based BATRAC + TTT training, or Lab-based Robot+ TTT.
- Home-based BATRAC Caregivers: An identified caregiver provided assistance as needed for the home-based intervention.
Period: Overall Study
Arm/Group | Home-based BATRAC | Lab-based BATRAC Plus TTT | Delayed Entry Usual Care | Home-based BATRAC Caregivers
Started | 11 | 9 | 9 | 19
Completed | 8 | 7 | 9 | 14
Not Completed | 3 | 2 | 0 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 5
Not completed — Adverse Event | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Caregivers did not receive outcome evaluations.
Groups:
- Home-based BATRAC: Home-based BATRAC training consisted of 60 minutes of training at home (45 minutes using the BATRAC and 15 minutes of TTT). BATRAC training included high intensity bilateral reaching and rest periods followed by 15 minutes of video guided transition to task training (TTT). The TTT videos were linked from the VA MyHealtheVet site to study specific Youtube videos of the study therapist demonstrating the exercise. Asynchronous communication between the therapist and participant was completed using the MyHealtheVet secure messaging system.
- Lab-based BATRAC Plus TTT: Lab-based BATRAC consisted of 60 minutes of training in the lab (45 minutes using BATRAC and 15 minutes of TTT). BATRAC training included high intensity bilateral reaching and rest periods followed by 15 minutes of therapist guided transition to task training (TTT).
- Delayed Entry Usual Care: Participants randomized to this group initially served as a control for the first 6 weeks of the study and did not receive any study interventions except the protocol study evaluations in the same time intervals as those receiving active interventions. They did received weekly phone calls to record general activity level. After serving as a control, this group entered into their randomized active intervention group of either lab-based BATRAC + TTT training, or Lab-based Robot+ TTT.
- Total: Total of all reporting groups
Arm/Group | Home-based BATRAC | Lab-based BATRAC Plus TTT | Delayed Entry Usual Care | Home-based BATRAC Caregivers | Total
Number analyzed (Participants) | 11 | 9 | 9 | 19 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.6) | 58.1 (10.6) | 58.7 (9.4) | 59.2 (17.1) | 60.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 11 | 24
  Male | 6 | 5 | 5 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 8 | 6 | 12 | 33
  White | 4 | 1 | 3 | 7 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 9 | 19 | 48
Wolf Motor Function Test Performance Time [Mean (Standard Deviation); unit: log (seconds)] — Each of the 15 tasks were timed to a maximum of 120 seconds. The mean WMFT time was log transformed to reduce the skewness of the values and a faster time (lower value) indicates a better outcome. Population: Caregivers did not receive outcome evaluations.
  log (seconds)
    number analyzed (Participants) | 11 | 9 | 9 | 0 | 29
    (all) | 3.2 (0.3) | 3.3 (0.4) | 3.2 (0.4) |  | 3.2 (0.4)
Fugl-Meyer [Mean (Standard Deviation); unit: units on a scale] — Scale ranging from 0-66 where a higher score indicates a better outcome. Population: Caregivers did not receive outcome evaluations.
  units on a scale
    number analyzed (Participants) | 11 | 9 | 9 | 0 | 29
    (all) | 32.3 (9.5) | 34.8 (12.1) | 32.2 (9.1) |  | 33 (9.9)
Stroke Impact Scale-hand domain [Mean (Standard Deviation); unit: units on a scale] — Scored on a 0-100 scale where a higher score indicates a better outcome. Population: Caregivers did not receive outcome evaluations.
  units on a scale
    number analyzed (Participants) | 11 | 9 | 9 | 0 | 29
    (all) | 28.2 (22.9) | 32.2 (35.7) | 40 (25.6) |  | 33.1 (27.7)

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test Performance Time (WMFT)
Description: The change between WMFT performance time from baseline to post-training was analyzed. Change = 6week WMFT log (time) minus baseline WMFT log (time). The WMFT performance time is a measure of movement speed to complete fifteen timed tasks up to a maximum of 120 seconds. A faster time (lower value) indicates a better outcome. The WMFT logarithm transformed time (WMFT log (time)) mean values were analyzed to reduce the skewness of the WMFT time values. The primary study outcome was the between group difference in the Home-based WMFT log (time) post-training compared to the control.
Time Frame: Final Training (week 6)
Population: Only 24 participants were included in the analysis, as we excluded patients who had no 6-week follow-up data on the primary outcome.
Measure: Mean (Standard Deviation); unit: log (seconds)
Groups:
- Home-Based BATRAC: Home-based BATRAC training consisted of 60 minutes of training at home (45 minutes using the BATRAC followed by 15 minutes of video guided transition to task training (TTT)). The BATRAC training included high intensity bilateral reaching and rest periods. The TTT videos were linked from the VA MyHealtheVet site to study specific Youtube videos of the study therapist demonstrating the exercise. Asynchronous communication between the therapist and participant was completed using the MyHealtheVet secure messaging system.
- Lab-based BATRAC Plus TTT: Lab-based BATRAC consisted of 60 minutes of training in the lab (45 minutes using BATRAC and 15 minutes of TTT). BATRAC training included high intensity bilateral reaching and rest periods followed by 15 minutes of therapist supervised and guided transition to task training (TTT).
- Delayed Entry Usual Care: Participants randomized to this group initially served as a control for the first 6 weeks of the study and did not receive any study interventions except for protocol study evaluations in the same time intervals as those receiving active interventions. They did receive weekly phone calls to record general activity level. After serving as a control, this group was entered into their randomized active intervention group of either lab-based BATRAC + TTT training, or Lab-based Robot+ TTT.
Arm/Group | Home-Based BATRAC | Lab-based BATRAC Plus TTT | Delayed Entry Usual Care
Number analyzed (Participants) | 8 | 7 | 9
log (seconds) | 3.6 (1.0) | 2.9 (1.2) | 3.1 (1.1)
Statistical Analysis 1: Comparison: Home-Based BATRAC vs Delayed Entry Usual Care; 78 participants were needed to generate a sample size of 22 per group and provide 80% power to detect a between group difference in mean Wolf time change (6 week - baseline) based on an a priori assumption of a mean change of 0 and 7.4 seconds respectively for the delayed entry usual care control and home-based BATRAC group; a SD of 7.6 and discontinuation rate of 15%; Test type: Superiority; p = 0.64, t-test, 2 sided — The primary analysis was a two sample t-test (alpha=0.05) of the mean WMFT log-time change at 6 weeks. The threshold for statistical significance was p-value = 0.05

2. Secondary Outcome: Fugl-Meyer Assessment Scale-Upper Extremity
Description: The Fugl-Meyer Assessment scale is a stroke specific motor impairment measure. It provides an assessment of graded volitional arm tasks and hand movements using a scale ranging from 0-66 where a higher score indicates a better outcome. It has been shown to be valid, reliable and have high inter-rater reliability and test/retest reliability.
Time Frame: Final Training (week 6)
Population: Only 24 participants completed the 6-week post-training evaluations and were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-Based BATRAC | Lab-based BATRAC Plus TTT | Delayed Entry Usual Care
Number analyzed (Participants) | 8 | 7 | 9
score on a scale | 32.3 (10.6) | 40.7 (13.5) | 32.0 (9.8)
Statistical Analysis 1: Comparison: Home-Based BATRAC vs Lab-based BATRAC Plus TTT vs Delayed Entry Usual Care; Within group changes from baseline to week 6 were assessed using analysis of variance; Test type: Superiority; p = 0.01, ANOVA — The lab-based group had significant within group mean Fugl-Meyer (FM) change at week 6; Dunnett's adjustments were used to compare the active intervention changes to the delayed-entry usual care control group
Statistical Analysis 2: Comparison: Home-Based BATRAC vs Delayed Entry Usual Care; FM change was analyzed using analysis of variance followed by Dunnett's adjustment for between group comparisons in the home-based BATRAC group compared to the delayed-entry control; Test type: Superiority; p = 0.97, ANOVA

3. Secondary Outcome: Stroke Impact Scale (SIS)-Hand Domain
Description: The Stroke Impact Scale is self-reported structured interview consisting of eight domains examining the physical, mental, and emotional changes that occur after a stroke and contribute to a change in quality of life. The SIS has been tested and found to be reliable, valid, and sensitive to change in the stroke population. It has four physical domains which assess strength, activities of daily living (ADL), mobility, and hand function abilities post stroke. These domains can be analyzed separately and scored on a 0-100 scale where a higher score indicates a better outcome.
Time Frame: Final Training (week 6)
Population: Only 24 participants completed the 6-week post-training evaluations and were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-Based BATRAC | Lab-based BATRAC Plus TTT | Delayed Entry Usual Care
Number analyzed (Participants) | 8 | 7 | 9
score on a scale | 31.9 (33.1) | 45.0 (26.5) | 39.4 (30.4)
Statistical Analysis 1: Comparison: Home-Based BATRAC vs Delayed Entry Usual Care; Within group SIS hand changes from baseline to week 6 were assessed using analysis of variance followed by comparisons to the delayed-entry usual care control using Dunnett's adjustment; Test type: Superiority; p = 0.31, ANOVA

ADVERSE EVENTS:
Time Frame: 14 to 20 weeks for each subject depending on randomization 14 weeks if randomized directly to intervention (6 weeks training + 8 weeks post training follow up). 20 weeks if randomized to delayed entry control (6 weeks control + 6 weeks training + 8 weeks post training).
Description: Adverse event reporting reflects the combined *total* number that received each intervention. Therefore, Home-Based BATRAC and Lab-Based BATRAC plus TTT listed below includes the delayed entry subject's AE's while randomized to each respective training group.
Groups:
- Delayed Entry Usual Care: Participants randomized to this group initially served as a control for the first 6 weeks of the study and did not receive any study interventions except the protocol study evaluations in the same time intervals as those receiving active interventions. They did receive weekly phone calls to record general activity level. After serving as a control, this group entered into their randomized active intervention group of either lab-based BATRAC + TTT training, or Lab-based Robot+ TTT.
Arm/Group | Home-based BATRAC | Lab-based BATRAC Plus TTT | Delayed Entry Usual Care | Home-based BATRAC Caregivers
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/9 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/9 | 0/19
Other Adverse Events (participants affected / at risk) | 4/15 | 4/14 | 1/9 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based BATRAC (N=15) | Lab-based BATRAC Plus TTT (N=14) | Delayed Entry Usual Care (N=9) | Home-based BATRAC Caregivers (N=19)
Fall at home (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — 1 subject sustained a finger fracture, 1 subject sustained a foot fracture and 1 subject denied injury but required medication change.
Dehydration and not taking medications (Social circumstances) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac Issues (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Sustained a back injury in motor vehicle accident on route to study appointment.
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Delayed onset muscle soreness

LIMITATIONS AND CAVEATS:
Previous VA guidance restricted MyHealtheVet (MHV) patient portal secure messaging (SM) from research making this study its first expansion as a tele-rehabilitation research tool. Several challenges related to equipment procurement and finalization of MHV patient portal research guidelines affected the recruitment timeline resulting in a small sample size. Therefore, the analysis of the primary outcome measure, a change from baseline to week 6 in Wolf performance time was underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT02665052/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT02665052/Prot_SAP_001.pdf